CLINICAL TRIAL: NCT02752451
Title: Cigar Box Arthroscopy: A Randomized Controlled Trial Validates Non-Anatomic Simulation Training of Novice Arthroscopy Skills
Brief Title: Cigar Box Arthroscopy: A Study of Non-Anatomic Arthroscopy Training
Acronym: CBA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1410543185
Record Dates: First submitted 2016-04-23; First posted 2016-04-27 (Estimated); Last update posted 2024-08-23 (Actual); Status verified 2016-06

CONDITIONS: Simulation Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- CO (Other): 8 subjects who did not undergo arthroscopy simulation training prior to assessment on cadaveric specimens. These served as controls.
  Interventions: Other: Pre-assesment education
- CBAT (Experimental): 8 Subjects who received 4 hours of simulation training on the Cigar Box Arthroscopy Trainer. They then underwent assessment on cadaveric specimens.
  Interventions: Other: Non-Anatomic Arthroscopy Simulation; Other: Pre-assesment education
- AKAT (Experimental): 8 Subjects who received 4 hours of simulation training on the Anatomic Knee Arthroscopy Trainer. They then underwent assessment on cadaveric specimens.
  Interventions: Other: Anatomic Arthroscopy Simulation; Other: Pre-assesment education

INTERVENTIONS:
Other: Non-Anatomic Arthroscopy Simulation — Knee arthroscopy training using Cigar Box Arthroscopy Trainer
  Arms: CBAT
Other: Anatomic Arthroscopy Simulation — Knee arthroscopy training using Anatomic Knee Arthroscopy Trainer
  Arms: AKAT
Other: Pre-assesment education — Reading material and lecture with only still images about performing diagnostic knee arthroscopy

SUMMARY:
Comparison of success rates of novice surgeons to attain proficiency in basic arthroscopy skills after receiving prior training with different simulation systems.

DETAILED DESCRIPTION:
A non-anatomic set of training modules utilizing cigar boxes was developed at our institution to instruct residents in the basics of knee arthroscopy. Twenty-four medical students with no prior arthroscopic or laparoscopic experience were enrolled as subjects. Sixteen subjects were randomized to participate in four hours of either the cigar box arthroscopy trainer (CBAT) or a previously validated anatomic knee arthroscopy trainer (AKAT). The remaining eight subjects served as controls (CO). All subjects underwent a one-hour formalized training session provided by our orthopaedic sports faculty. Subjects' skills were assessed by one of two faculty members through repeated attempts at performing a diagnostic knee arthroscopy on a cadaveric specimen. Objective scores were given using the Basic Arthroscopic Knee Skill Scoring System. Total cost differences were also calculated.

ELIGIBILITY:
Inclusion Criteria:

* First or Second year medical student with no prior arthroscopy or laparoscopy training.

Exclusion Criteria:

* Having previously received education in arthroscopy or laparoscopy or handled these instruments.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Success rate in reaching a level of minimum proficiency | 1 hour
  Subjects were told to perform serial knee arthroscopic examinations on a cadaveric specimen over one hour. Evaluators used a validated objective scoring system to assess performance and which subjects were able to attain a level of minimum proficiency.

SECONDARY OUTCOMES:
Number of attempts to reach minimum proficiency | 1 Hour

IPD SHARING:
Plan to Share IPD: Undecided